CLINICAL TRIAL: NCT02944383
Title: A 12-Week, Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy Safety and Tolerability of Gemcabene in Subjects With Severe Hypertriglyceridemia (INDIGO-1)
Brief Title: A 12-Week Study to Assess the Efficacy Safety and Tolerability of Gemcabene in Subjects With Severe Hypertriglyceridemia
Acronym: INDIGO-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroBo Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GEM-401
Record Dates: First submitted 2016-10-24; First posted 2016-10-25 (Estimated); Results first posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Severe Hypertriglyceridemia; Mixed Dyslipidaemia
Keywords: Hypertriglycerides
MeSH Terms: conditions — Hypertriglyceridemia | interventions — gemcabene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gemcabene 300 mg (Experimental): Participants received 300 mg Gemcabene orally, once daily for 12 weeks.
  Interventions: Drug: Gemcabene
- Gemcabene 600 mg (Experimental): Participants received 600 mg Gemcabene orally, once daily for 12 weeks.
  Interventions: Drug: Gemcabene
- Placebo (Placebo Comparator): Participants received matching placebo orally, once daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gemcabene — Gemcabene tablets administered orally once daily, for 12 weeks.
  Arms: Gemcabene 300 mg; Gemcabene 600 mg
Drug: Placebo — Placebo tablets administered orally once daily, for 12 weeks.
  Arms: Placebo

SUMMARY:
A 12-Week, Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy Safety and Tolerability of Gemcabene in Subjects with Severe Hypertriglyceridemia (INDIGO-1)

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria will be eligible to participate in the study:

1. Provision of written and signed informed consent (by subject or legal guardian) prior to any study-specific procedure;
2. Male or female (neither pregnant or lactating) ≥18 years of age at time of consent;

   1. Women of child-bearing potential must have a negative serum pregnancy test at the Screening Visit and negative urine dipstick on Study Day 1 prior to dosing in order to qualify for the study. Women who are surgically sterile or are clinically confirmed to be post-menopausal (i.e., documented amenorrhea for ≥ 1 year in the absence of other biological or physiological causes) are not considered to be of child-bearing potential;
   2. Women of child-bearing potential must agree to use acceptable methods of contraception throughout the duration of the study and for 30 days after the last dose of study drug. For this study, double-barrier contraception is required.
3. Currently on a self-reported, stable, low-fat, low-cholesterol diet in combination with stable statins with or without ezetimibe (10 mg QD) for at least 12 weeks prior to the Screening Visit;
4. Mean fasting TG value ≥ 500 mg/dL to < 1500 mg/dL (with the higher value no more than 50% greater than the lower value) from the S1 and S2 Visits (or alternatively S2 and S3);
5. Physical examination, including vital signs, that is within normal limits or clinically acceptable to the Investigator;
6. Weight ≥ 50 kg; with a body mass index (BMI) ≤ 45 kg/m²; and
7. Subjects with Type 2 diabetes who take anti-diabetes pharmacologic therapy must be on a stable a regimen for at least 3 months, with no planned changes in medications for the study duration.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from participation in the study:

1. Known and previously documented homozygous genetic deficiencies (LPL, ApoC-II, ApoC-III, ApoA-V, GPIHBP1, or LMF1);
2. History of pancreatitis within the last 6 months prior to screening (Visit S1);
3. History of bariatric surgery; symptomatic gallstone disease, unless treated with cholecystectomy;
4. Abnormal liver function test at the Pre-Screening Visit or any of the Screening Visits (aspartate aminotransferase or alanine aminotransferase > 2 × the upper limit of normal [ULN], total bilirubin > 1.5 × ULN, or alkaline phosphatase > 2 × ULN based on appropriate age and gender normal values). Subjects with bilirubin > 1.5 × ULN and history of Gilbert's syndrome may be included; reflexive direct bilirubin testing will be used to confirm Gilbert's syndrome;
5. Active liver disease (e.g., cirrhosis, alcoholic liver disease, hepatitis B [HBV], hepatitis C [HCV], autoimmune hepatitis, liver failure, liver cancer), history of liver transplant, known diagnosis of human immunodeficiency virus (HIV), or acquired immune deficiency virus;
6. Moderate to severe renal insufficiency defined as an estimated GFR < 60 mL/min/1.73 m2 (calculated using The Chronic Kidney Disease Epidemiology Collaboration equation) at the Pre-Screening Visit or at any of the Screening Visits;
7. Abnormal urinalysis (proteinuria greater than trace or any male or non-menstruating female with greater than trace hematuria), confirmed by reflexive urine protein:creatinine ratio testing;
8. Uncontrolled thyroid disease: hyperthyroidism or hypothyroidism as defined by thyroid stimulating hormone (TSH) below the lower limit of normal or > 1.5 × ULN, respectively, based on results from the Pre-Screening Visit or the Screening Visit. If controlled, treatment should be stable for at least 3 months prior to the Screening Visit;
9. Type 1 diabetes mellitus or uncontrolled type 2 diabetes mellitus HbA1c value ≥8.5% based on results from the Pre-Screening Visit or the Screening Visit), or any diabetic subject taking a thiazolidinedione (e.g., pioglitazone, rosiglitazone);
10. New York Heart Association Class III or IV heart failure (see Appendix C);
11. Myocardial infarction, severe or unstable angina pectoris, coronary angioplasty, coronary artery bypass graft, or other major cardiovascular events resulting in hospitalization within 3 months of the Screening Visit (S1). Subjects with adequately treated stable angina, per Investigator assessment, may be included;
12. Uncontrolled cardiac arrhythmia or prolonged QT on the Screening Visit or Study Day 1 prior to dosing ECG (QTcF > 450 msec for men and >470 msec for women) or known family history of prolonged QT or unexplained sudden cardiac death;
13. Uncontrolled hypertension, defined as sitting systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg, and confirmed by repeat measurement;
14. Currently receiving cancer treatment(s) or, in the Investigator's opinion, at risk of relapse for recent cancer;
15. Inadequate washout of a PCSK9 inhibitor (8 weeks prior to the Screening Visit S1), a fibrate lipid lowering agent (6 weeks prior to the Screening Visit S1), niacin > 200 mg/day, OMG-3, bile acid sequestrants or other lipid lowering therapies (4 weeks prior to the Screening Visit S1);
16. Use of any excluded medications or supplements within 3 months prior to S1 (e.g., potent cytochrome P450 [CYP] 3A4 inhibitors, see Appendix D);
17. Hypersensitivity to or a history of significant adverse reactions to any fibrate lipid regulating agent;
18. History of drug or alcohol abuse within the past year or inability to comply with protocol requirements, including subject alcohol restrictions (see Section 5.6.3);
19. Previously treated with gemcabene (i.e., CI-1027); participation in another clinical study of an investigational agent or device concurrently or within 1 month prior to the Screening Visit, or use of an investigational agent within 1 month or 5 half-lives (if known), whichever is longer, prior to the Screening Visit; or
20. Any other finding which, in the opinion of the Investigator, would compromise the subject's safety or participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2016-12; Primary Completion 2018-01-11 (Actual); Study Completion 2018-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Golden, MD, Study Director — NeuroBo Pharmaceuticals Inc.
Locations (49):
- United States (48):
  - Appalachian Research Associates, Fort Payne, Alabama
  - Del Sol Research Mangagement, LLC, Tucson, Arizona
  - Westside Medical Associates of Los Angeles, Beverly Hills, California
  - Hope Clinical Research, Canoga Park, California
  - SC Clinical Research, Garden Grove, California
  - National Research Institute, Huntington Park, California
  - National Research Institute, Los Angeles, California
  - Paradigm Clinical Research, San Diego, California
  - Paradigm Research, Wheat Ridge, Colorado
  - Excel Medical Research, Boca Raton, Florida
  - Meridien Research, Bradenton, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Indago Research and Health Center, Hialeah, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Sunrise Medical Research, Lauderdale Lakes, Florida
  - San Marcus Research Clinic, Inc., Miami, Florida
  - Millenium Clinical Research, Inc., Miami, Florida
  - Medcare Research, Miami, Florida
  - AR Developoment Solutions, Miami Lakes, Florida
  - Soma Medical Research, West Palm Beach, Florida
  - Evanston Premier Clinical Research, Evanston, Illinois
  - Midwest Institute for Clinical Research, Inc., Indianapolis, Indiana
  - Richard Lochamy, M.D., Junction City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Clinical Trials Management, LLC, Covington, Louisiana
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Elite Clinical Research, Jackson, Mississippi
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - CHEAR Center, LLC, The Bronx, New York
  - Advantage Clinical Trials, The Bronx, New York
  - Eastern Carolina Medical Clinic, Benson, North Carolina
  - Physicians East, NA, Farmville, North Carolina
  - Physicians East, NA, Greenville, North Carolina
  - Cary Medical Clinic, Morrisville, North Carolina
  - Optimed Research, Columbus, Ohio
  - PriMed Clinical Research, Dayton, Ohio
  - Green and Seidner Family Practice Associates, Lansdale, Pennsylvania
  - BTC of Lincoln, Lincoln, Rhode Island
  - Carolinas Research Partners, LLC, Rock Hill, South Carolina
  - Airline Complete Healthcare, Houston, Texas
  - Sante Clinical Research, Kerrville, Texas
  - FMC Science, Lampasas, Texas
  - Clinical Investigations of Texas, Plano, Texas
  - Sun Research Institute, San Antonio, Texas
  - Clinical Investigation Specialists, Kenosha, Wisconsin
- Ecogene-21, Chicoutimi, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcabene 600 mg: Participants received 600 milligram (mg) Gemcabene orally, once daily for 12 weeks.
Period: Overall Study
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Started | 30 | 30 | 31
Completed | 29 | 30 | 30
Not Completed | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All randomized participants who received at least 1 dose of study drug and had at least 1 post-baseline efficacy assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 31 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (9.10) | 51.5 (9.50) | 54.6 (12.06) | 54.1 (10.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 12 | 18
  Male | 25 | 29 | 19 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 13 | 10 | 35
  Not Hispanic or Latino | 18 | 17 | 21 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 2 | 4
  White | 28 | 29 | 25 | 82
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 2
Triglycerides [TG] [Median (Full Range); unit: Milligram per deciliter (mg/dL)] | 637 [456.7 to 1477.7] | 641.17 [387.0 to 1658.7] | 658.33 [442.0 to 1205.7] | 643.0 [387.0 to 1658.7]
Non-high-density lipoprotein cholesterol (non-HDL-C) [Median (Full Range); unit: mg/dL] | 238.75 [121.5 to 324.5] | 190.0 [104.0 to 448.5] | 201.00 [80.5 to 373.5] | 205.00 [80.5 to 448.5]
High-density lipoprotein cholesterol (HDL-C) [Median (Full Range); unit: mg/dL] | 28.50 [17.0 to 46.0] | 28.00 [19.0 to 39.0] | 29.00 [17.0 to 56.0] | 28.0 [17.0 to 56.0]
Very low-density lipoprotein cholesterol (VLDL-C) [Median (Full Range); unit: mg/dL] | 108.50 [54.0 to 230.0] | 102.50 [27.0 to 359.0] | 117.00 [51.0 to 350.0] | 110.00 [27.0 to 359.0]
Total Cholesterol (TC) [Median (Full Range); unit: mg/dL] | 273.00 [138.5 to 352.5] | 219.00 [131.0 to 487.5] | 235.00 [103.5 to 401.5] | 237.00 [103.5 to 487.5]
Low-density lipoprotein cholesterol (LDL-C) [Median (Full Range); unit: mg/dL] | 97.00 [39.0 to 233.0] | 87.00 [31.0 to 183.0] | 76.00 [17.0 to 197.0] | 87.00 [17.0 to 233.0]
High-density lipoprotein Triglyceride (HDL-TG) [Median (Full Range); unit: mg/dL] | 34.5 [21 to 180] | 33.0 [22 to 122] | 36.0 [15 to 97] | 35.0 [15 to 180]
Very low-density lipoprotein Triglyceride (VLDL-TG) [Median (Full Range); unit: mg/dL] | 476.0 [232 to 1757] | 462.0 [83 to 3384] | 541.0 [217 to 1602] | 506.0 [83 to 3384]
Low-density lipoprotein Triglyceride (LDL-TG) [Median (Full Range); unit: mg/dL] | 59.0 [15 to 99] | 47.5 [26 to 104] | 54.0 [26 to 82] | 53.0 [15 to 104]
Apolipoprotein B (ApoB) [Median (Full Range); unit: mg/dL] | 113.5 [66 to 186] | 107.0 [64 to 186] | 110.0 [44 to 157] | 111.0 [44 to 186]
Apolipoprotein A-I (ApoA-I) [Median (Full Range); unit: mg/dL] | 130.0 [101 to 168] | 121.0 [84 to 175] | 133.0 [100 to 194] | 130.0 [84 to 194]
Apolipoprotein A-II (ApoA-II) [Median (Full Range); unit: mg/dL] | 35.0 [25 to 46] | 33.0 [25 to 46] | 34.0 [23 to 55] | 34.0 [23 to 55]
Apolipoprotein C-II (ApoC-II) [Median (Full Range); unit: mg/dL] — Population: FAS Population. Here, number analyzed signifies participants with available data.
  mg/dL
    number analyzed (Participants) | 30 | 29 | 30 | 89
    (all) | 10 [4 to 10] | 10 [1 to 10] | 10 [5 to 10] | 10 [1 to 10]
Apolipoprotein C-III (ApoC-III) [Median (Full Range); unit: mg/dL] | 25.5 [9 to 60] | 25.0 [6 to 59] | 27.0 [8 to 57] | 26.0 [6 to 60]
Apolipoprotein B (ApoE) [Median (Full Range); unit: mg/dL] | 8.1 [4 to 22] | 7.8 [3 to 29] | 9.1 [3 to 32] | 8.5 [3 to 32]
High-sensitivity C-reactive protein (hsCRP) [Median (Full Range); unit: mg/dL] | 3.65 [0.6 to 10.5] | 2.75 [0.4 to 64.1] | 2.50 [0.2 to 13.6] | 3.20 [0.2 to 64.1]
Fibrinogen [Median (Full Range); unit: mg/dL] | 418.5 [343 to 572] | 415.0 [279 to 1020] | 375.0 [243 to 753] | 400.0 [243 to 1020]
Adiponectin [Median (Full Range); unit: Microgram per milliliter (μg/mL)] | 3.9 [2 to 9] | 4.3 [1 to 9] | 4.4 [2 to 20] | 4.2 [1 to 20]
Serum amyloid A [Median (Full Range); unit: Milligram per Liter (mg/L)] | 5.9 [2 to 36] | 4.8 [1 to 196] | 5.0 [1 to 29] | 5.3 [1 to 196]
Interleukin-6 [Median (Full Range); unit: Picogram per milliliter (pg/mL)] — Population: FAS Population. Here, number analyzed signifies participants with available data.
  Picogram per milliliter (pg/mL)
    number analyzed (Participants) | 29 | 30 | 31 | 90
    (all) | 2.6 [1 to 8] | 2.1 [1 to 20] | 2.5 [1 to 20] | 2.3 [1 to 20]
Angiopoietin 4 [Median (Full Range); unit: Nanogram per milliliter (ng/mL)] | 204.1 [116 to 315] | 171.8 [99 to 345] | 165.7 [87 to 404] | 176.6 [87 to 404]
Lipoprotein size [Median (Full Range); unit: Nanometer (nm)] — Particle size for VLDL, HDL, LDL were reported. Population: FAS Population. Here, number analyzed signifies participants with available data.
  Nanometer (nm)
    Very low density lipoprotein (VLDL) | 64.90 [44.4 to 82.7] | 62.25 [47.8 to 85.6] | 68.80 [40.1 to 79.5] | 64.60 [40.1 to 85.6]
    low density lipoprotein (LDL): number analyzed (Participants) | 30 | 30 | 29 | 89
    low density lipoprotein (LDL) | 19.60 [19.4 to 21.7] | 19.60 [19.3 to 21.0] | 19.60 [19.3 to 21.6] | 19.60 [19.3 to 21.7]
    High density lipoprotein (HDL) | 8.700 [7.80 to 9.10] | 8.500 [7.90 to 9.30] | 8.700 [7.90 to 9.60] | 8.700 [7.80 to 9.60]
HDL Particle Number [Median (Full Range); unit: Micro mole per Liter (umol/L)] | 30.450 [18.10 to 39.00] | 28.500 [19.10 to 47.10] | 30.800 [18.80 to 48.40] | 29.700 [18.10 to 48.40]
Lipoprotein Particle Number [Median (Full Range); unit: Nano mole per Liter (nmol/L)]
  VLDL and Chylomicron Particles | 147.90 [34.6 to 289.8] | 145.35 [17.9 to 357.4] | 140.90 [36.0 to 325.9] | 147.20 [17.9 to 357.4]
  LDL Particles | 1447.50 [593.0 to 2969.0] | 1228.50 [457.0 to 2946.0] | 1178.00 [214.0 to 2460.0] | 1259.00 [214.0 to 2969.0]
  Intermediate Density Lipoprotein (IDL) Particles | 164.5 [8 to 570] | 114.0 [1 to 988] | 137.0 [3 to 466] | 137.0 [1 to 988]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to End of Study (EOS) in Fasting Serum Triglycerides (TG)
Description: EOS was defined as the average of the week 10 and week 12 values. If either the week 10 or week 12 value was missing, then the single value (week 10 or week 12) was used. Completely missing values (both week 10 and week 12) were imputed using last observation carried forward (LOCF).
Time Frame: Baseline, EOS (average of week 10 and 12)
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Groups:
- Gemcabene 300 mg: Participants received 300 mg of Gemcabene orally, once daily for 12 weeks.
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 31
Percent Change | -47.32 [-59.58 to -30.93] | -32.95 [-48.53 to -12.21] | -27.30 [-41.90 to 10.12]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Test type: Superiority; p = 0.0063, Ranked ANCOVA; Randomized treatment group & randomized baseline statin (yes or no) are included as factors, & outcome (ranked) at baseline is included as covariate; Median Difference (Net) = -19.02, 95% CI 2-sided [-33.07 to -4.25] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Test type: Superiority; p = 0.2350, Ranked ANCOVA; [statistical method as in outcome 1, analysis 1]; Median Difference (Net) = -7.63, 95% CI 2-sided [-25.88 to 7.05] — Estimates generated from Hodges-Lehmann method

2. Secondary Outcome: Percent Change From Baseline in Fasting Serum TG
Time Frame: Baseline, Weeks 2, 6, 10 and 12
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 31
Percent Change
  Week 2 | -27.46 [-49.03 to -14.03] | -27.10 [-46.77 to 2.24] | -27.07 [-37.53 to 11.01]
  Week 6 | -38.63 [-50.24 to -18.99] | -25.11 [-46.46 to -5.47] | -22.18 [-41.48 to -5.17]
  Week 10 | -49.90 [-58.32 to -25.53] | -32.83 [-47.65 to -18.99] | -18.75 [-46.07 to 11.55]
  Week 12 | -41.88 [-57.53 to -25.04] | -36.01 [-48.92 to -10.10] | -37.30 [-48.35 to -5.46]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 2; Test type: Other; p = 0.1663, Ranked ANCOVA — Ranked ANCOVA results are obtained using a model where the outcome is ranked, randomized treatment group and randomized baseline statin (yes or no) are included as factors, and outcome (ranked) at baseline is included as a covariate
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 2; Test type: Superiority; p = 0.6195, Ranked ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 6; Test type: Superiority; p = 0.0436, Ranked ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 6; Test type: Superiority; p = 0.5000, Ranked ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0007, Ranked ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.1161, Ranked ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.1830, Ranked ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.8762, Ranked ANCOVA — [p-value comment as in outcome 2, analysis 1]

3. Secondary Outcome: Change From Baseline in Fasting Serum TG
Description: EOS was defined as the average of the week 10 and week 12 values. If either the week 10 or week 12 value was missing, then the single value (week 10 or week 12) was used. Completely missing values (both week 10 and week 12) were imputed using LOCF.
Time Frame: Baseline, Weeks 2, 6, 10, 12 and EOS (average of week 10 and 12)
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Groups:
- Gemcabene 600 mg: Participants received 600 mg of Gemcabene orally, once daily for 12 weeks.
- Placebo: Participants received 300 mg of Gemcabene orally, once daily for 12 weeks.
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 31
mg/dL
  Week 2 | -221.83 [-359.00 to -83.67] | -161.00 [-306.67 to 11.67] | -163.67 [-302.67 to 58.00]
  Week 6 | -272.33 [-355.33 to -162.67] | -173.83 [-301.33 to -27.67] | -130.00 [-263.67 to -33.0]
  Week 10 | -298.33 [-456.33 to -141.00] | -173.50 [-390.67 to -105.67] | -131.00 [-312.67 to 91.00]
  Week 12 | -234.33 [-482.33 to -165.00] | -230.67 [-308.33 to -59.67] | -202.67 [-407.67 to -32.00]
  EOS | -288.42 [-411.83 to -156.33] | -219.67 [-340.83 to -71.17] | -154.00 [-380.33 to 49.83]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 2; Test type: Superiority; p = 0.1780, Ranked ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 2; Test type: Superiority; p = 0.7615, Ranked ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 6; Test type: Superiority; p = 0.0162, Ranked ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 6; Test type: Superiority; p = 0.3710, Ranked ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0010, Ranked ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0988, Ranked ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.2594, Ranked ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.9099, Ranked ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0219, Ranked ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.3494, Ranked ANCOVA — [p-value comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percent Change From Baseline in TC
Description: as for outcome 3
Time Frame: Baseline, Weeks 2, 6, 10, 12 and EOS (average of week 10 and 12)
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 31
Percent Change
  Week 2 | -12.67 [-24.84 to 2.33] | -4.48 [-20.00 to 4.73] | -2.67 [-14.74 to 7.38]
  Week 6 | -17.00 [-26.25 to 0.85] | -8.68 [-13.66 to 4.67] | -6.12 [-13.43 to 5.31]
  Week 10 | -17.23 [-30.86 to -6.50] | -8.44 [-17.83 to 2.29] | -2.42 [-12.56 to 10.20]
  Week 12 | -10.25 [-30.94 to -1.81] | -8.62 [-13.18 to 7.34] | -6.93 [-18.18 to 14.97]
  EOS | -13.65 [-31.91 to -5.13] | -7.28 [-19.92 to 6.49] | -2.82 [-16.46 to 10.80]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 2; Test type: Superiority; p = 0.0391, Ranked ANCOVA — Results are obtained using a model where outcome is ranked, randomized treatment group, randomized baseline statin (yes or no), & randomized qualifying TG stratum are included as factors, & outcome (ranked) at baseline is included as a covariate
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 2; Test type: Superiority; p = 0.2455, Ranked ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 6; Test type: Superiority; p = 0.0260, Ranked ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 6; Test type: Superiority; p = 0.5704, Ranked ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0009, Ranked ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0846, Ranked ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.1763, Ranked ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.5576, Ranked ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 9: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0086, Ranked ANCOVA — [p-value comment as in outcome 4, analysis 1]; Median Difference (Net) = -14.66, 95% CI 2-sided [-24.68 to -4.39] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 10: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.1516, Ranked ANCOVA — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Net) = -5.06, 95% CI 2-sided [-15.02 to 3.64] — Estimates generated from Hodges-Lehmann method

5. Secondary Outcome: Change From Baseline in TC
Description: as for outcome 3
Time Frame: Baseline, Weeks 2, 6, 10, 12 and EOS (average of week 10 and 12)
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 31
mg/dL
  Week 2 | -25.75 [-65.00 to 5.00] | -10.25 [-51.50 to 8.00] | -5.50 [-36.00 to 17.00]
  Week 6 | -41.50 [-76.50 to 2.00] | -18.75 [-32.50 to 7.00] | -13.50 [-31.50 to 6.50]
  Week 10 | -41.25 [-89.00 to -13.50] | -16.00 [-49.50 to 3.00] | -2.50 [-33.50 to 20.50]
  Week 12 | -28.25 [-79.00 to -3.50] | -19.75 [-53.50 to 14.00] | -14.00 [-42.50 to 29.50]
  EOS | -35.50 [-90.50 to -13.50] | -14.25 [-51.50 to 8.50] | -3.00 [-36.50 to 25.00]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 2; Test type: Superiority; p = 0.0386, Ranked ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 2; Test type: Superiority; p = 0.1206, Ranked ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 6; Test type: Superiority; p = 0.0364, Ranked ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 6; Test type: Superiority; p = 0.4312, Ranked ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0010, Ranked ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0407, Ranked ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.1433, Ranked ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.2866, Ranked ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 9: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0056, Ranked ANCOVA — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 10: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0789, Ranked ANCOVA — [p-value comment as in outcome 4, analysis 1]

6. Secondary Outcome: Percent Change From Baseline in Non-HDL-C
Description: as for outcome 3
Time Frame: Baseline, Weeks 2, 6, 10, 12 and EOS (average of week 10 and 12)
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 31
Percent Change
  Week 2 | -13.92 [-29.92 to -0.78] | -6.35 [-21.52 to 3.23] | -3.29 [-15.62 to 8.90]
  Week 6 | -22.57 [-32.16 to -0.77] | -10.55 [-14.29 to 2.84] | -7.77 [-16.28 to 4.23]
  Week 10 | -22.18 [-35.66 to -7.92] | -11.18 [-22.19 to 2.23] | -7.66 [-17.18 to 13.36]
  Week 12 | -13.31 [-36.34 to -3.37] | -9.92 [-19.31 to 11.35] | -10.56 [-22.62 to 19.21]
  EOS | -15.64 [-38.11 to -5.26] | -12.01 [-21.88 to 7.10] | -3.98 [-20.80 to 11.56]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 2; Test type: Superiority; p = 0.0277, Ranked ANCOVA — Results are obtained using a model where the outcome is ranked, randomized treatment group, randomized baseline statin (yes or no), & randomized qualifying TG stratum are included as factors, & outcome (ranked) at baseline is included as a covariate
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 2; Test type: Superiority; p = 0.2502, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 6; Test type: Superiority; p = 0.0161, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 6; Test type: Superiority; p = 0.6567, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0010, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.1257, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.1440, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.7642, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 9: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0107, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -16.40, 95% CI 2-sided [-28.31 to -4.51] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 10: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.2466, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -5.32, 95% CI 2-sided [-16.73 to 5.52] — Estimates generated from Hodges-Lehmann method

7. Secondary Outcome: Change From Baseline in Non-HDL-C
Description: as for outcome 3
Time Frame: Baseline, Weeks 2, 6, 10, 12 and EOS (average of week 10 and 12)
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 31
mg/dL
  Week 2 | -30.75 [-73.50 to -2.00] | -12.25 [-52.50 to 5.50] | -6.50 [-36.00 to 15.00]
  Week 6 | -43.50 [-81.50 to -2.50] | -19.75 [-34.50 to 5.00] | -16.50 [-38.50 to 6.00]
  Week 10 | -45.00 [-93.00 to -15.50] | -23.00 [-52.00 to 4.00] | -7.50 [-39.50 to 22.00]
  Week 12 | -29.00 [-90.00 to -9.00] | -22.25 [-54.50 to 15.00] | -16.00 [-51.00 to 31.00]
  EOS | -36.50 [-93.00 to -14.50] | -21.25 [-50.00 to 11.50] | -7.00 [-42.50 to 21.50]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 2; Test type: Superiority; p = 0.0211, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 2; Test type: Superiority; p = 0.1304, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 6; Test type: Superiority; p = 0.0318, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 6; Test type: Superiority; p = 0.4607, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0012, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0592, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.1170, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.3138, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 9: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0090, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 10: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.1317, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

8. Secondary Outcome: Percent Change From Baseline in VLDL-C
Description: as for outcome 3
Time Frame: Baseline, Weeks 2, 6, 10, 12 and EOS (average of week 10 and 12)
Population: FAS Population. Missing values were imputed by LOCF. Here, Number analyzed signifies those participants who were evaluable at each specified time point only.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 31
Percent Change
  Week 2: number analyzed (Participants) | 12 | 11 | 9
  Week 2 | -46.19 [-57.52 to -21.18] | -46.27 [-63.78 to -5.41] | -29.59 [-48.36 to 18.87]
  Week 6: number analyzed (Participants) | 18 | 13 | 16
  Week 6 | -36.41 [-50.00 to -18.75] | -43.31 [-50.51 to -4.55] | -33.50 [-53.68 to -2.57]
  Week 10: number analyzed (Participants) | 30 | 27 | 30
  Week 10 | -32.71 [-60.00 to -14.41] | -16.67 [-52.90 to 11.01] | -7.85 [-41.03 to 28.93]
  Week 12 | -31.34 [-51.74 to -6.92] | -19.14 [-39.80 to 15.38] | -31.69 [-44.21 to 20.57]
  EOS | -31.95 [-50.00 to -12.50] | -15.95 [-50.51 to 15.38] | -17.57 [-39.89 to 27.71]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 2; Test type: Superiority; p = 0.2395, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 2; Test type: Superiority; p = 0.6380, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 6; Test type: Superiority; p = 0.7468, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 6; Test type: Superiority; p = 0.8483, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0008, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0938, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.3201, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.9010, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 9: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0156, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -19.31, 95% CI 2-sided [-39.06 to -1.49] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 10: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.3456, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -5.98, 95% CI 2-sided [-28.51 to 17.26] — Estimates generated from Hodges-Lehmann method

9. Secondary Outcome: Change From Baseline in VLDL-C
Description: as for outcome 3
Time Frame: Baseline, Weeks 2, 6, 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 31
mg/dL
  Week 2: number analyzed (Participants) | 12 | 11 | 9
  Week 2 | -47.00 [-74.00 to -18.50] | -60 [-84.00 to -4.00] | -29.00 [-59.00 to 10.00]
  Week 6: number analyzed (Participants) | 18 | 13 | 16
  Week 6 | -37.50 [-57.00 to -12.00] | -50.00 [-70.00 to -3.00] | -31.50 [-67.50 to -1.50]
  Week 10: number analyzed (Participants) | 30 | 27 | 30
  Week 10 | -25.50 [-73.00 to -17.00] | -15.00 [-68.00 to 12.00] | -7.00 [-48.00 to 20.00]
  Week 12 | -26.00 [-68.00 to -10.00] | -19.00 [-73.00 to 12.00] | -24.00 [-62.00 to 21.00]
  EOS | -32.50 [-56.00 to -10.50] | -13.00 [-71.50 to 12.00] | -19.50 [-63.00 to 23.00]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 2; Test type: Superiority; p = 0.3714, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 2; Test type: Superiority; p = 0.4415, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 6; Test type: Superiority; p = 0.7902, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 6; Test type: Superiority; p = 0.6999, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0015, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0796, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.4225, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.7687, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 9: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0437, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 10: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.2735, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

10. Secondary Outcome: Percent Change From Baseline in HDL-C
Description: as for outcome 3
Time Frame: Baseline, Weeks 2, 6, 10, 12 and EOS (average of week 10 and 12)
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 31
Percent Change
  Week 2 | 5.96 [-3.03 to 28.57] | 3.85 [-7.14 to 14.29] | 4.35 [-7.69 to 15.38]
  Week 6 | 5.33 [-6.67 to 17.65] | 7.42 [-7.14 to 13.33] | 0.00 [-3.70 to 21.21]
  Week 10 | 5.87 [-4.35 to 29.41] | 7.14 [-4.00 to 18.75] | 10.34 [0.00 to 22.22]
  Week 12 | 14.72 [-9.52 to 23.81] | 7.29 [-3.70 to 20.00] | 7.69 [-4.35 to 25.00]
  EOS | 9.30 [-7.50 to 23.53] | 7.04 [-7.69 to 17.86] | 8.70 [-3.85 to 21.74]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 2; Test type: Superiority; p = 0.1042, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 2; Test type: Superiority; p = 0.6204, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 6; Test type: Superiority; p = 0.8659, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 6; Test type: Superiority; p = 0.9658, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.8238, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.4874, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.9467, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.7467, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 9: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.9081, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -0.41, 95% CI 2-sided [-10.77 to 10.75] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 10: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.5480, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -2.38, 95% CI 2-sided [-11.82 to 6.86] — Estimates generated from Hodges-Lehmann method

11. Secondary Outcome: Change From Baseline in HDL-C
Description: as for outcome 3
Time Frame: Baseline, Weeks 2, 6, 10, 12 and EOS (average of week 10 and 12)
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 31
mg/dL
  Week 2 | 2.00 [-1.00 to 7.00] | 1.00 [-2.00 to 4.00] | 1 [-3.00 to 4.00]
  Week 6 | 1.50 [-2.00 to 5.00] | 2.00 [-2.00 to 4.00] | 0.00 [-1.00 to 6.00]
  Week 10 | 2.00 [-1.00 to 7.00] | 2.00 [-1.00 to 4.00] | 3.00 [0.00 to 5.00]
  Week 12 | 4.00 [-3.00 to 8.00] | 2.00 [-1.00 to 5.00] | 2.00 [-1.00 to 8.00]
  EOS | 3.00 [-2.00 to 6.00] | 2.00 [-2.00 to 4.00] | 2.00 [-1.00 to 5.00]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 2; Test type: Superiority; p = 0.1485, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 2; Test type: Superiority; p = 0.6008, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 6; Test type: Superiority; p = 0.9409, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 6; Test type: Superiority; p = 0.9292, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.8455, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.5256, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 7: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.9217, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 8: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.7401, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 9: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.9386, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 10: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.6352, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

12. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
Percent Change
  Week 10: number analyzed (Participants) | 29 | 27 | 29
  Week 10 | -10.5 [-28.1 to 4.3] | -2.7 [-9.2 to 5.6] | 0.0 [-5.1 to 8.9]
  Week 12 | -4.7 [-26.1 to 6.6] | 0.5 [-8.6 to 16.2] | 4.8 [-6.4 to 13.0]
  EOS | -5.9 [-25.7 to 4.9] | -1.9 [-8.7 to 11.4] | 2.8 [-5.0 to 7.6]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0165, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.3075, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.1069, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.6101, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0351, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -12.04, 95% CI 2-sided [-23.79 to -1.08] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.3746, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -3.15, 95% CI 2-sided [-9.86 to 4.25] — Estimates generated from Hodges-Lehmann method

13. Secondary Outcome: Change From Baseline in Apolipoprotein B
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: FAS Population. Missing values were imputed by LOCF. Here, overall number of participants analyzed (N) signifies those participants who were evaluable for this outcome measure and number analyzed signifies those participants who were evaluable at each specified time point only.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
mg/dL
  Week 10: number analyzed (Participants) | 29 | 27 | 29
  Week 10 | -10.0 [-37.0 to 4.0] | -4.0 [-13.0 to 6.0] | 0.0 [-5.0 to 9.0]
  Week 12 | -7.0 [-30.0 to 8.0] | 0.5 [-13.0 to 12.0] | 5.5 [-6.0 to 16.0]
  EOS | -8.5 [-34.5 to 5.5] | -1.8 [-13.0 to 9.5] | 2.8 [-5.5 to 9.0]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0133, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.2044, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0855, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.5114, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0289, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.2950, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

14. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-I
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
Percent Change
  Week 10: number analyzed (Participants) | 29 | 27 | 29
  Week 10 | -3.3 [-9.7 to 6.3] | 5.1 [-5.6 to 12.2] | 2.7 [-3.4 to 6.5]
  Week 12 | 5.9 [-4.9 to 12.1] | 4.0 [-2.7 to 13.2] | 2.1 [-3.6 to 10.8]
  EOS | 1.2 [-4.5 to 8.1] | 4.6 [-1.4 to 12.4] | 2.0 [-5.4 to 9.9]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.1992, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.9945, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.5139, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.8085, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.7644, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -0.77, 95% CI 2-sided [-6.31 to 4.85] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.9499, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Net) = 1.33, 95% CI 2-sided [-4.34 to 6.66] — Estimates generated from Hodges-Lehmann method

15. Secondary Outcome: Change From Baseline in Apolipoprotein A-I
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
mg/dL
  Week 10: number analyzed (Participants) | 29 | 27 | 29
  Week 10 | 5.0 [-13 to 7] | 6.0 [-7.0 to 13.0] | 4.0 [-5.0 to 9.0]
  Week 12 | 8.0 [-6.0 to 16.0] | 4.5 [-3.0 to 15.0] | 2.5 [-4.0 to 15.0]
  EOS | 1.5 [-7.0 to 10.0] | 5.5 [-2.0 to 13.0] | 2.5 [-7.0 to 14.0]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.1521, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.8982, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.6228, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.9622, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.6643, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.9071, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

16. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-II
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
Percent Change
  Week 10: number analyzed (Participants) | 29 | 27 | 29
  Week 10 | -3.2 [-8.1 to 5.9] | 6.9 [-3.3 to 12.5] | 0.0 [-7.1 to 7.3]
  Week 12 | 0.0 [-2.9 to 10.0] | 4.5 [0.0 to 15.2] | 0.0 [-6.9 to 7.5]
  EOS | 0.0 [-5.4 to 5.6] | 5.3 [-3.1 to 12.1] | 0.0 [-5.6 to 8.1]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.5647, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.1073, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.3858, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0916, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.9473, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = 0.0, 95% CI 2-sided [-5.56 to 5.26] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0911, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = 4.54, 95% CI 2-sided [-1.83 to 9.95] — Estimates generated from Hodges-Lehmann method

17. Secondary Outcome: Change From Baseline in Apolipoprotein A-II
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
mg/dL
  Week 10: number analyzed (Participants) | 29 | 27 | 29
  Week 10 | -1.0 [-3.0 to 2.0] | 2.0 [-1.0 to 4.0] | 0.0 [-2.0 to 3.0]
  Week 12 | 0.0 [-1.0 to 4.0] | 1.5 [0.0 to 5.0] | 0.0 [-2.0 to 3.0]
  EOS | 0.0 [-1.5 to 2.0] | 1.8 [-1.0 to 4.0] | 0.0 [-2.0 to 2.5]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.4623, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.1678, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.4390, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.1290, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.9627, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0911, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

18. Secondary Outcome: Percent Change From Baseline in Apolipoprotein C-II
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 29
Percent Change
  Week 10: number analyzed (Participants) | 29 | 27 | 27
  Week 10 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Week 12 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [-10.0 to 0.0]
  EOS | 0.0 [-5.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [-5.6 to 0.0]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.2882, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.4474, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.7875, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0600, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.9832, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = 0.00, 95% CI 2-sided [0.00 to 0.00] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.1352, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = 0.00, 95% CI 2-sided [0.00 to 0.00] — Estimates generated from Hodges-Lehmann method

19. Secondary Outcome: Change From Baseline in Apolipoprotein C-II
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 29
mg/dL
  Week 10: number analyzed (Participants) | 29 | 27 | 27
  Week 10 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Week 12 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [-1.0 to 0.0]
  EOS | 0.0 [-0.5 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [-0.5 to 0.0]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.2857, ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.4486, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.7640, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0560, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.9954, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.1298, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

20. Secondary Outcome: Percent Change From Baseline in Apolipoprotein C-III
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
Percent Change
  Week 10: number analyzed (Participants) | 29 | 27 | 28
  Week 10 | -21.1 [-40.0 to -4.7] | -14.3 [-35.6 to 11.1] | -3.6 [-33.2 to 16.5]
  Week 12 | -17.6 [-35.5 to -5.6] | -6.4 [-27.7 to 14.3] | -10.7 [-37.5 to 0.0]
  EOS | -17.6 [-39.6 to -7.1] | -11.3 [-31.5 to 8.3] | -8.1 [-29.3 to 9.1]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0161, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.1806, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.2657, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.5996, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0270, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -11.39, 95% CI 2-sided [-28.81 to 2.08] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.5263, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -0.92, 95% CI 2-sided [-16.88 to 15.50] — Estimates generated from Hodges-Lehmann method

21. Secondary Outcome: Change From Baseline in Apolipoprotein C-III
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
mg/dL
  Week 10: number analyzed (Participants) | 29 | 27 | 28
  Week 10 | -6.0 [-12.0 to -2.0] | -4.0 [-9.0 to 1.0] | -1.0 [-10.5 to 3.0]
  Week 12 | -4.0 [-9.0 to -1.0] | -2.0 [-6.0 to 2.0] | -3.0 [-13.0 to 0.0]
  EOS | -5.5 [-12.0 to -2.0] | -3.3 [-8.0 to 2.0] | -2.0 [-9.5 to 2.0]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0345, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.2709, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.3255, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.7391, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0808, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.6509, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

22. Secondary Outcome: Percent Change From Baseline in Apolipoprotein E
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
Percent Change
  Week 10: number analyzed (Participants) | 29 | 27 | 29
  Week 10 | -36.3 [-46.4 to -26.4] | -22.6 [-42.4 to 8.2] | -9.2 [-39.0 to 14.3]
  Week 12 | -27.5 [-43.5 to -1.6] | -14.6 [-41.7 to 10.0] | -25.7 [-43.4 to 14.7]
  EOS | -33.2 [-45.3 to -13.5] | -16.7 [-43.1 to 10.6] | -10.4 [-40.2 to 20.0]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0004, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0412, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.1937, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.4740, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0116, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -14.32, 95% CI 2-sided [-34.13 to 3.89] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.1109, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -3.66, 95% CI 2-sided [-23.85 to 14.26] — Estimates generated from Hodges-Lehmann method

23. Secondary Outcome: Change From Baseline in Apolipoprotein E
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
mg/dL
  Week 10: number analyzed (Participants) | 29 | 27 | 29
  Week 10 | -3.0 [-5.4 to -1.9] | -1.8 [-4.2 to 0.5] | -0.9 [-4.4 to 1.0]
  Week 12 | -2.2 [-4.0 to -0.1] | -1.4 [-4.1 to 0.7] | -1.8 [-5.5 to 1.6]
  EOS | -2.9 [-4.9 to -1.0] | -1.3 [-4.2 to 0.5] | -0.9 [-4.9 to 1.5]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0002, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0161, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.3043, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.4639, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0210, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0992, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

24. Secondary Outcome: Percent Change From Baseline in LDL-C
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
Percent Change
  Week 10: number analyzed (Participants) | 29 | 26 | 29
  Week 10 | -13.64 [-27.03 to 26.32] | 4.39 [-14.00 to 29.03] | 0.00 [-7.92 to 32.14]
  Week 12 | -7.94 [-26.39 to 22.97] | 5.20 [-13.04 to 26.67] | 25.43 [2.99 to 42.86]
  EOS | -13.36 [-25.79 to 19.66] | 5.26 [-12.68 to 27.94] | 14.73 [0.00 to 37.50]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.1512, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.8400, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0244, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.1803, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0307, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -24.41, 95% CI 2-sided [-42.73 to -9.94] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.5326, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -8.73, 95% CI 2-sided [-23.33 to 7.68] — Estimates generated from Hodges-Lehmann method

25. Secondary Outcome: Change From Baseline in LDL-C
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
mg/dL
  Week 10: number analyzed (Participants) | 29 | 26 | 29
  Week 10 | -12.00 [-42.00 to 15.00] | 3.00 [-14.00 to 23.00] | 0.00 [-6.0 to 18.00]
  Week 12 | -10.00 [-23.00 to 17] | 4.50 [-16.00 to 25.00] | 17.50 [2.00 to 29.00]
  EOS | -11.50 [-31.00 to 19.00] | 5.75 [-11.50 to 21.00] | 8.75 [0.00 to 20.50]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.1705, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.9193, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0224, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.2387, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0600, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.6878, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

26. Secondary Outcome: Percent Change From Baseline in LDL-TG
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
Percent Change
  Week 10: number analyzed (Participants) | 29 | 26 | 28
  Week 10 | -17.1 [-35.6 to -4.2] | -12.2 [-33.3 to 7.1] | 0.8 [-19.8 to 13.9]
  Week 12 | -17.5 [-45.8 to 9.1] | -7.2 [-28.6 to 31.0] | -6.0 [-18.6 to 12.7]
  EOS | -20.0 [-37.5 to 4.4] | -9.3 [-17.8 to 16.1] | -6.8 [-16.7 to 13.6]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0298, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0196, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.2219, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.4078, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0605, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -15.34, 95% CI 2-sided [-31.68 to 1.30] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.1768, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -4.08, 95% CI 2-sided [-19.91 to 7.32] — Estimates generated from Hodges-Lehmann method

27. Secondary Outcome: Change From Baseline in LDL-TG
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
mg/dL
  Week 10: number analyzed (Participants) | 29 | 26 | 28
  Week 10 | -11.0 [-21.0 to -1.0] | -6.5 [-19.0 to 2.0] | 0.5 [-10.0 to 7.5]
  Week 12 | -10.0 [-29.0 to 4.0] | -4.0 [-11.0 to 10.0] | -3.0 [-11.0 to 7.0]
  EOS | -12.5 [-25.0 to 2.0] | -4.0 [-12.0 to 5.0] | -3.3 [-8.5 to 8.5]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0084, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0047, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.1574, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.3235, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0367, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0948, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

28. Secondary Outcome: Percent Change From Baseline in VLDL-TG
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
Percent Change
  Week 10: number analyzed (Participants) | 29 | 26 | 29
  Week 10 | -39.7 [-60.6 to -21.2] | -32.8 [-58.6 to 28.7] | -11.0 [-53.9 to 19.5]
  Week 12 | -34.8 [-59.0 to -15.3] | -27.0 [-47.5 to 8.8] | -37.3 [-56.4 to -6.9]
  EOS | -35.2 [-57.7 to -23.3] | -30.8 [-52.8 to 38.4] | -23.9 [-51.3 to 10.6]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0037, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.1328, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.4364, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.8129, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0347, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -15.29, 95% CI 2-sided [-36.54 to 2.35] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.3617, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -2.14, 95% CI 2-sided [-25.78 to 23.62] — Estimates generated from Hodges-Lehmann method

29. Secondary Outcome: Change From Baseline in VLDL-TG
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: FAS Population. Missing values were imputed by LOCF. Here, overall number of participants analyzed (N) signifies those participants who were evaluable for this outcome measure and number analyzed signifies those participants who were evaluable at specified time point only.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
mg/dL
  Week 10: number analyzed (Participants) | 29 | 26 | 29
  Week 10 | -170.0 [-493.0 to -86.0] | -129.5 [-241.0 to 84.0] | -77.0 [-274.0 to 67.0]
  Week 12 | -139.0 [-351.0 to -83.0] | -103.5 [-320.0 to 52.0] | -193.5 [-524.0 to -28.0]
  EOS | -164.0 [-468.0 to -76.5] | -116.5 [-373.0 to 71.5] | -126.8 [-384.0 to 92.0]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0085, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.2112, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.7301, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.6283, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0919, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.5497, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

30. Secondary Outcome: Percent Change From Baseline in HDL-TG
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 31
Percent Change
  Week 10 | -27.5 [-51.6 to -11.8] | -6.5 [-35.8 to 11.5] | -6.1 [-26.7 to 19.2]
  Week 12 | -23.9 [-54.1 to 3.0] | -17.3 [-37.8 to -2.9] | -11.1 [-31.3 to 21.7]
  EOS | -20.6 [-52.7 to 3.4] | -11.2 [-39.0 to 3.8] | -1.4 [-29.3 to 26.7]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0009, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0351, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.1561, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0268, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0516, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -22.30, 95% CI 2-sided [-42.96 to -1.67] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 6: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0125, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -13.06, 95% CI 2-sided [-32.83 to 4.88] — Estimates generated from Hodges-Lehmann method

31. Secondary Outcome: Change From Baseline in HDL-TG
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 31
mg/dL
  Week 10 | -8.0 [-25.0 to -3.0] | -2.0 [-15.0 to 3.0] | -2.0 [-11.0 to 6.0]
  Week 12 | -8.0 [-25.0 to 1.0] | -5.5 [-17.0 to -1.0] | -4.0 [-12.0 to 5.0]
  EOS | -7.0 [-25.0 to 1.0] | -3.5 [-16.0 to 1.0] | -0.5 [-10.0 to 6.0]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0023, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0356, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.2284, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0213, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0330, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0221, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

32. Secondary Outcome: Percent Change From Baseline in Lipoprotein Size
Description: Percent change from baseline in Particle size for VLDL, HDL and LDL were reported.
Time Frame: Baseline, Week 12
Population: FAS Population. Missing values were imputed by LOCF. Here, overall number of participants analyzed (N) signifies those participants who were evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 29 | 29
Percent Change
  VLDL | -7.83 [-16.46 to -0.31] | -6.36 [-14.90 to 9.72] | -5.17 [-16.55 to 3.34]
  LDL | 0.00 [0.00 to 1.52] | 0.00 [0.00 to 0.95] | 0.51 [-0.51 to 1.03]
  HDL | 0.000 [-2.299 to 2.273] | 0.000 [-2.353 to 2.353] | 0.000 [-2.151 to 1.205]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; VLDL; Test type: Superiority; p = 0.2632, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -2.67, 95% CI 2-sided [-10.17 to 5.67] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; VLDL; Test type: Superiority; p = 0.5382, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = 2.02, 95% CI 2-sided [-6.77 to 9.71] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; LDL; Test type: Superiority; p = 0.1727, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = 0.00, 95% CI 2-sided [-0.51 to 1.01] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; LDL; Test type: Superiority; p = 0.4567, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = 0.00, 95% CI 2-sided [-0.51 to 0.51] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; HDL; Test type: Superiority; p = 0.6142, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = 0.00, 95% CI 2-sided [-1.21 to 1.47] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; HDL; Test type: Superiority; p = 0.2409, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -0.02, 95% CI 2-sided [-2.23 to 1.29] — Estimates generated from Hodges-Lehmann method

33. Secondary Outcome: Change From Baseline in Lipoprotein Size
Description: Change from baseline in Particle size for VLDL, HDL and LDL were reported.
Time Frame: Baseline, Week 12
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: nm
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 29 | 29
nm
  VLDL | -5.10 [-10.60 to -0.20] | -3.90 [-10.80 to 5.90] | -3.10 [-12.20 to 2.30]
  LDL | 0.00 [0.00 to 0.30] | 0.00 [0.00 to 0.20] | 0.10 [-0.10 to 0.20]
  HDL | 0.000 [-0.200 to 0.200] | 0.000 [-0.200 to 0.200] | 0.000 [-0.200 to 0.100]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; VLDL; Test type: Superiority; p = 0.2721, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; VLDL; Test type: Superiority; p = 0.5669, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; LDL; Test type: Superiority; p = 0.1686, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; LDL; Test type: Superiority; p = 0.4308, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; HDL; Test type: Superiority; p = 0.5495, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; HDL; Test type: Superiority; p = 0.2384, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

34. Secondary Outcome: Percent Change From Baseline in Lipoprotein Particle Number
Description: Percent change from baseline in particle number for VLDL & chylomicron, LDL and IDL were reported.
Time Frame: Baseline, Week 12
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 29 | 29
Percent Change
  VLDL and Chylomicron Particles | -15.82 [-22.82 to 7.60] | -3.88 [-19.10 to 23.25] | -4.03 [-14.33 to 26.67]
  LDL Particles | -9.83 [-32.15 to 7.53] | -10.20 [-25.14 to 15.54] | 13.96 [-13.73 to 36.46]
  IDL Particles | -73.1 [-90.1 to 17.9] | -2.2 [-83.2 to 36.3] | 16.7 [-67.5 to 217.6]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; VLDL & Chylomicron particles; Test type: Superiority; p = 0.0781, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -13.99, 95% CI 2-sided [-33.76 to 2.55] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; VLDL & Chylomicron particles; Test type: Superiority; p = 0.9901, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -2.10, 95% CI 2-sided [-19.36 to 19.01] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; LDL Particles; Test type: Superiority; p = 0.0717, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -25.23, 95% CI 2-sided [-43.62 to -5.10] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; LDL Particles; Test type: Superiority; p = 0.1548, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -16.09, 95% CI 2-sided [-36.78 to 3.76] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; IDL Particles; Test type: Superiority; p = 0.0428, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -47.16, 95% CI 2-sided [-119.58 to -5.78] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; IDL Particles; Test type: Superiority; p = 0.1836, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -26.13, 95% CI 2-sided [-121.44 to 19.48] — Estimates generated from Hodges-Lehmann method

35. Secondary Outcome: Change From Baseline in Lipoprotein Particle Number
Description: Change from baseline in particle number for VLDL & chylomicron, LDL and IDL were reported.
Time Frame: Baseline, Week 12
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 29 | 29
nmol/L
  VLDL and Chylomicron Particles | -10.90 [-49.10 to 10.50] | -6.40 [-32.30 to 24.50] | -4.30 [-27.30 to 32.30]
  IDL Particles | -67.0 [-191.0 to 24.0] | -14.0 [-72.0 to 31.0] | 1.0 [-96.0 to 86.0]
  LDL Particles | -103.00 [-525.00 to 88.00] | -82.00 [-341.00 to 160.00] | 160.0 [-134.0 to 425]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; VLDL & Chylomicron Particles; Test type: Superiority; p = 0.1251, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; VLDL & Chylomicron Particles; Test type: Superiority; p = 0.9047, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; LDL Particles; Test type: Superiority; p = 0.0788, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; LDL Particles; Test type: Superiority; p = 0.1222, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; IDL Particles; Test type: Superiority; p = 0.0734, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; IDL Particles; Test type: Superiority; p = 0.4210, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

36. Secondary Outcome: Percent Change From Baseline in HDL Particle Number
Time Frame: Baseline, Week 12
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 29 | 29
Percent Change | -0.578 [-11.111 to 13.889] | 0.304 [-5.079 to 12.253] | 0.000 [-5.296 to 8.696]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Test type: Superiority; p = 0.9672, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = 0.43, 95% CI 2-sided [-8.12 to 9.07] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Test type: Superiority; p = 0.7993, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = 1.58, 95% CI 2-sided [-5.31 to 8.69] — Estimates generated from Hodges-Lehmann method

37. Secondary Outcome: Change From Baseline in HDL Particle Number
Time Frame: Baseline, Week 12
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 29 | 29
umol/L | -0.200 [-4.100 to 3.400] | 0.100 [-1.600 to 3.800] | 0.000 [-1.600 to 2.300]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Test type: Superiority; p = 0.8602, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Test type: Superiority; p = 0.8555, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

38. Secondary Outcome: Percent Change From Baseline in High-sensitivity C-reactive Protein
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
Percent Change
  Week 10: number analyzed (Participants) | 29 | 27 | 29
  Week 10 | -33.33 [-54.29 to 0.00] | -26.67 [-44.90 to 15.56] | -10.00 [-30.00 to 14.29]
  Week 12 | -16.67 [-60.61 to 0.00] | -25.48 [-57.89 to 5.56] | 10.99 [-28.57 to 42.86]
  EOS | -23.68 [-53.57 to 3.45] | -16.94 [-55.26 to 17.11] | -0.71 [-25.00 to 50.00]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0583, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.2289, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0416, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0150, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0718, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -26.21, 95% CI 2-sided [-54.29 to -1.26] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.1248, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -18.68, 95% CI 2-sided [-50.00 to 7.31] — Estimates generated from Hodges-Lehmann method

39. Secondary Outcome: Change From Baseline in High-sensitivity C-reactive Protein
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
mg/dL
  Week 10: number analyzed (Participants) | 29 | 27 | 29
  Week 10 | -0.90 [-1.90 to 0.00] | -0.40 [-1.50 to 0.20] | -0.10 [-1.20 to 0.20]
  Week 12 | -0.60 [-2.00 to 0.00] | -0.50 [-1.50 to 0.10] | 0.10 [-0.40 to 1.20]
  EOS | -0.75 [-1.95 to 0.10] | -0.28 [-1.50 to 0.40] | -0.02 [-0.60 to 0.65]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.2397, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.5399, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0409, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0073, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0976, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.1899, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

40. Secondary Outcome: Percent Change From Baseline in Fibrinogen
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
Percent Change
  Week 10: number analyzed (Participants) | 29 | 25 | 29
  Week 10 | 1.2 [-11.0 to 13.5] | -6.7 [-14.2 to 7.4] | -3.5 [-10.2 to 8.8]
  Week 12 | -1.8 [-15.0 to 5.4] | -11.4 [-19.3 to 0.8] | -3.4 [-11.6 to 4.6]
  EOS | -0.2 [-13.5 to 8.9] | -8.4 [-15.1 to 0.8] | -3.1 [-9.6 to 6.8]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.1747, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.4576, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.1549, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.2427, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.1379, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = 1.51, 95% CI 2-sided [-6.26 to 8.73] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.2490, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -6.02, 95% CI 2-sided [-13.10 to 0.51] — Estimates generated from Hodges-Lehmann method

41. Secondary Outcome: Change From Baseline in Fibrinogen
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
mg/dL
  Week 10: number analyzed (Participants) | 29 | 25 | 29
  Week 10 | 5.0 [-50.0 to 54.0] | -22.0 [-53.0 to 26.0] | -15.0 [-38.0 to 37.0]
  Week 12 | -7.0 [-63.0 to 23.0] | -50.0 [-80.0 to 3.0] | -12.0 [-46.0 to 17.0]
  EOS | -1.0 [-56.5 to 40.5] | -35.0 [-71.0 to 3.0] | -14.3 [-36.5 to 22.5]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.1550, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.6604, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0952, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.3006, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0642, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.3185, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

42. Secondary Outcome: Percent Change From Baseline in Serum Amyloid A
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
Percent Change
  Week 10: number analyzed (Participants) | 29 | 27 | 29
  Week 10 | -33.3 [-45.8 to -16.2] | -19.2 [-38.2 to -3.0] | -12.5 [-31.5 to 0.0]
  Week 12 | -36.7 [-58.7 to -15.4] | -29.2 [-58.6 to 0.0] | -7.2 [-20.6 to 17.3]
  EOS | -31.8 [-51.1 to -1.7] | -19.6 [-52.9 to 8.9] | -7.2 [-21.7 to 11.3]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0679, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.4126, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0095, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0172, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0359, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -23.23, 95% CI 2-sided [-41.54 to -3.64] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0812, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -16.06, 95% CI 2-sided [-38.62 to 5.61] — Estimates generated from Hodges-Lehmann method

43. Secondary Outcome: Change From Baseline in Serum Amyloid A
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 30
mg/L
  Week 10: number analyzed (Participants) | 29 | 27 | 29
  Week 10 | -1.5 [-2.5 to -0.7] | -0.6 [-2.1 to -0.1] | -0.4 [-1.6 to 0.0]
  Week 12 | -2.1 [-3.3 to -0.6] | -0.9 [-2.7 to 0.0] | -0.3 [-1.3 to 0.9]
  EOS | -1.5 [-2.7 to -0.1] | -0.8 [-2.7 to 0.5] | -0.2 [-1.1 to 0.6]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.1362, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.6458, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0209, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0822, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0504, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.1315, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

44. Secondary Outcome: Percent Change From Baseline in Adiponectin
Description: as for outcome 3
Time Frame: Baseline, Week 12 and EOS (average of week 10 and 12)
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 29 | 30
Percent Change
  Week 12 | 12.9 [0.9 to 36.5] | 12.4 [-6.5 to 31.6] | 1.2 [-12.7 to 15.1]
  EOS | 12.9 [0.9 to 36.5] | 12.4 [-6.5 to 31.6] | 1.2 [-12.7 to 15.1]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0843, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.3587, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0843, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = 12.99, 95% CI 2-sided [-0.54 to 25.51] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.3587, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = 7.98, 95% CI 2-sided [-3.70 to 21.39] — Estimates generated from Hodges-Lehmann method

45. Secondary Outcome: Change From Baseline in Adiponectin
Description: as for outcome 3
Time Frame: Baseline, Week 12 and EOS (average of week 10 and 12)
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: μg/mL
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 29 | 30
μg/mL
  Week 12 | 0.3 [0.0 to 0.9] | 0.3 [-0.2 to 0.8] | 0.0 [-0.7 to 0.6]
  EOS | 0.3 [0.0 to 0.9] | 0.3 [-0.2 to 0.8] | 0.0 [-0.7 to 0.6]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0768, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.4346, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0768, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.4346, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

46. Secondary Outcome: Percent Change From Baseline in Angiopoietin 4
Description: as for outcome 3
Time Frame: Baseline, Week 12 and EOS (average of week 10 and 12)
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 29 | 30
Percent Change
  Week 12 | 8.5 [-5.1 to 21.7] | -1.6 [-18.6 to 20.8] | 1.1 [-6.9 to 15.2]
  EOS | 8.5 [-15.1 to 21.7] | -1.6 [-18.6 to 20.8] | 1.1 [-6.9 to 15.2]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.5411, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.2574, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.5411, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = 3.11, 95% CI 2-sided [-9.59 to 14.86] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.2574, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -7.31, 95% CI 2-sided [-19.30 to 5.76] — Estimates generated from Hodges-Lehmann method

47. Secondary Outcome: Change From Baseline in Angiopoietin 4
Description: as for outcome 3
Time Frame: Baseline, Week 12 and EOS (average of week 10 and 12)
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 29 | 30
ng/mL
  Week 12 | 15.7 [-14.1 to 56.7] | -2.0 [-36.8 to 48.5] | 2.8 [-9.1 to 22.5]
  EOS | 15.7 [-14.1 to 56.7] | -2.0 [-36.8 to 48.5] | 2.8 [-9.1 to 22.5]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.3998, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.3659, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.3998, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.3659, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

48. Secondary Outcome: Percent Change From Baseline in Interleukin-6
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 29
Percent Change
  Week 10: number analyzed (Participants) | 28 | 25 | 28
  Week 10 | -7.7 [-22.7 to 34.0] | -10.2 [-37.3 to 14.7] | -1.1 [-31.6 to 49.1]
  Week 12 | -6.2 [-21.7 to 41.6] | -7.5 [-34.4 to 21.3] | -10.6 [-27.2 to 1.2]
  EOS | -5.3 [-17.7 to 30.7] | -4.8 [-28.3 to 37.4] | -4.2 [-27.2 to 35.5]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.8823, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.3788, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.1091, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.6867, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.3156, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = 9.07, 95% CI 2-sided [-12.22 to 36.34] — Estimates generated from Hodges-Lehmann method
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.9734, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]; Median Difference (Net) = -0.30, 95% CI 2-sided [-24.58 to 25.43] — Estimates generated from Hodges-Lehmann method

49. Secondary Outcome: Change From Baseline in Interleukin-6
Description: as for outcome 3
Time Frame: Baseline, Weeks 10, 12 and EOS (average of week 10 and 12)
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 29 | 30 | 29
pg/mL
  Week 10: number analyzed (Participants) | 28 | 25 | 28
  Week 10 | -0.1 [-0.7 to 0.4] | -0.1 [-0.8 to 0.3] | -0.0 [-0.9 to 1.0]
  Week 12 | -0.1 [-0.6 to 0.7] | -0.2 [-0.7 to 0.3] | -0.2 [-0.5 to 0.0]
  EOS | -0.1 [-0.6 to 0.6] | -0.2 [-0.7 to 0.4] | -0.1 [-0.6 to 0.4]
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.9772, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.5213, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.1582, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.4588, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.4264, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.8107, Ranked ANCOVA — [p-value comment as in outcome 6, analysis 1]

50. Secondary Outcome: Percentage of Participants Achieving a TG Value < 500 mg/dL (5.65 mmol/L)
Description: as for outcome 3
Time Frame: Weeks 10, 12 and EOS (average of week 10 and 12)
Population: FAS Population. Missing values were imputed by LOCF.
Measure: Number; unit: Percentage of participants
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
Number analyzed (Participants) | 30 | 30 | 31
Percentage of participants
  Week 10 | 73.3 | 63.3 | 41.9
  Week 12 | 63.3 | 53.3 | 41.9
  EOS | 66.7 | 56.7 | 45.2
Statistical Analysis 1: Comparison: Gemcabene 600 mg vs Placebo; Week 10; Test type: Superiority; p = 0.0093, Regression, Logistic — Logistic regression results are obtained using a model with randomized treatment group, randomized baseline statin (yes or no), and baseline TG value as independent factors; Odds Ratio (OR) = 5.38, 95% CI 2-sided [1.51 to 19.08] — The OR is an estimate of the odds of achieving a TG value < 500 mg/dL associated with the corresponding Gemcabene group relative to the placebo group at a given visit
Statistical Analysis 2: Comparison: Gemcabene 300 mg vs Placebo; Week 10; Test type: Superiority; p = 0.1070, Regression, Logistic — [p-value comment as in outcome 50, analysis 1]; Odds Ratio (OR) = 2.57, 95% CI 2-sided [0.82 to 8.07] — [estimate comment as in outcome 50, analysis 1]
Statistical Analysis 3: Comparison: Gemcabene 600 mg vs Placebo; Week 12; Test type: Superiority; p = 0.0865, Regression, Logistic — [p-value comment as in outcome 50, analysis 1]; Odds Ratio (OR) = 2.57, 95% CI 2-sided [0.87 to 7.53]
Statistical Analysis 4: Comparison: Gemcabene 300 mg vs Placebo; Week 12; Test type: Superiority; p = 0.3990, Regression, Logistic — [p-value comment as in outcome 50, analysis 1]; Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.55 to 4.48] — [estimate comment as in outcome 50, analysis 1]
Statistical Analysis 5: Comparison: Gemcabene 600 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.0772, Regression, Logistic — [p-value comment as in outcome 50, analysis 1]; Odds Ratio (OR) = 2.75, 95% CI 2-sided [0.90 to 8.42] — [estimate comment as in outcome 50, analysis 1]
Statistical Analysis 6: Comparison: Gemcabene 300 mg vs Placebo; EOS (average of week 10 and 12); Test type: Superiority; p = 0.4315, Regression, Logistic — [p-value comment as in outcome 50, analysis 1]; Odds Ratio (OR) = 1.54, 95% CI 2-sided [0.53 to 4.48] — [estimate comment as in outcome 50, analysis 1]

ADVERSE EVENTS:
Time Frame: Baseline to End of study (up to Day 113)
Arm/Group | Gemcabene 600 mg | Gemcabene 300 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 1/31
Other Adverse Events (participants affected / at risk) | 16/30 | 14/30 | 20/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcabene 600 mg (N=30) | Gemcabene 300 mg (N=30) | Placebo (N=31)
Cystitis (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Gemcabene 600 mg (N=30) | Gemcabene 300 mg (N=30) | Placebo (N=31)
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 4
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 3
Nasopharyngitis (Infections and infestations) | 1 | 0 | 2
Sinusitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract Infection (Infections and infestations) | 0 | 1 | 2
Influenza (Infections and infestations) | 0 | 1 | 1
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 0/5 | 0/1 | 1/12 — Gender specific event, total number adjusted to female participants.
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 1 | 0
Haemoglobin decreased (Investigations) | 2 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 0 | 0
Haematocrit decreased (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0
Urine analysis abnormal (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0
Immunology test abnormal (Investigations) | 0 | 0 | 1
Hyperinsulinaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Breast cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/5 | 0/1 | 1/12 — Gender specific event, total number adjusted to female participants.
Headache (Nervous system disorders) | 1 | 1 | 2
Cervical radiculopathy (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Nephropathy toxic (Renal and urinary disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1/5 | 0/1 | 0/12 — Gender specific event, total number adjusted to female participants.
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1/5 | 0/1 | 0/12 — Gender specific event, total number adjusted to female participants.
Breast mass (Reproductive system and breast disorders) | 0/5 | 0/1 | 1/12 — Gender specific event, total number adjusted to female participants.
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin tightness (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT02944383/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/83/NCT02944383/SAP_001.pdf